CLINICAL TRIAL: NCT04303026
Title: A Randomized Placebo Controlled Trial Testing The Effect of Zoledronic Acid on Hip Osteoarthritis
Brief Title: The Effect of Zoledronic Acid on Patients With Osteoarthritis of the Hip
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Hormone Laboratory, Aker University Hospital, Oslo, Norway (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Morten Halkjær Iversen, Principal investigator, Vestre Viken Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018030; 2019-000757-31 (EudraCT Number)
Record Dates: First submitted 2020-03-02; First posted 2020-03-10 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Zoledronic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 70 participants are allocated randomly to either treatment group or placebo group by a member not part of the study group through an internet based website (Studyrandomizer.com) Participants cannot cross over, but they can withdraw from the study or treatment/Placebo or request alternate treatment (surgery)
Who Masked: Participant, Care Provider, Investigator
Masking Description: The treatment and placebo is administered through an infusion. Both will be administered in an identical infusion bag and are colorless. The mixing is performed by the same person who randomizes, less than 24 hours before administration. The bags are then put in a refrigerator and picked up later by a study nurse for administration. There is no "personal contact".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): Participants receiving active treatment with two infusions of Zoledronic Acid 5 mg with 3 months interval mixed in 100 ml 0.9% saline
  Interventions: Drug: Zoledronic Acid
- Placebo Group (Placebo Comparator): Participants receiving Placebo with two infusions of 100 ml 0.9% saline with 3 months interval.
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Zoledronic Acid — 5mg IV infusion
  Other Names: Active Treatment
  Arms: Treatment Group
Drug: Saline 0.9% — Placebo Group. Saline 0.9% 100 ml infusion
  Other Names: Placebo
  Arms: Placebo Group

SUMMARY:
Hip Osteoarthritis (OA) is one of the most common diseases affecting the ageing population. No specific and safe treatment slowing the development of hip OA as reflected in reduced joint space narrowing has been developed so far. Implantation of hip prosthesis has been a great success, but is expensive and puts a great financial pressure on hospitals and national healthcare programs. It also poses risks of serious complications. Current non-surgical treatment options focus on pain management and physiotherapy.

Bisphosphonates have been shown to exert multiple beneficial effects in OA. Animal studies have demonstrated that bisphosphonates protect against subchondral bone degradation and preserve articular cartilage in mice and rats with OA.

In this study 70 participants will be treated with either Zoledronic Acid (a potent Bisphosphonate) or Placebo (Saltwater). Allocation will be random and both parties are blinded. The investigators hypothesis is that participants treated with Zoledronic acid will have less pain, and better function after 12 months. The results will be tested with functional and pain scores, and functional tests. The study team will also measure the effects on disease related quality of life, bone quality measurements and the effect on bone marrow lesions on MRI (magnetic resonance imaging) and histological examination

DETAILED DESCRIPTION:
Background Hip Osteoarthritis (OA) is one of the most common diseases affecting the ageing population. No specific and safe treatment slowing the development of hip OA as reflected in reduced joint space narrowing has been developed so far. Implantation of hip prosthesis has been a great success, but is expensive and puts a great financial pressure on hospitals and national healthcare programs. It also poses risks of serious complications. Current non-surgical treatment options focus on pain management and physiotherapy.

Bisphosphonates have been shown to exert multiple beneficial effects in OA, not only through effects on subchondral bone, but also through chondroprotection and possibly by inhibiting synovitis. Animal studies have demonstrated that bisphosphonates protect against subchondral bone degradation and preserve articular cartilage in mice and rats with OA. Efforts to further improve subchondral bone using a combination of zoledronic acid (ZA) and parathyroid hormone (PTH), was, however, shown to be ineffective.

Rationale for study Effects of bisphosphonates in OA

Bisphosphonates may target Pain and OA development by several different mechanisms:

Anti-osteoclastic action:

Increased bone turnover in OA causes bone loss and osteoporosis of subchondral bone beneath the thickened subchondral plate, which alters flexibility, and increases the risk of microfracture, which may cause of bone marrow lesions (BMLs) in OA. Bisphosphonates may also increase the strength of subchondral bone by reducing turnover and improve bone material properties.

Osteoclasts mediate the extension of channels from marrow spaces into the non-calcified articular cartilage. This leads to loss of integrity at the osteochondral junction exposing subchondral nerves to proinflammatory and pain inducing factors from the synovial fluid. This action has also been shown to induce sensory nerve growth into the non-calcified articular cartilage.

Osteoclasts may also reduce pH at the osteochondral junction, thereby sensitizing and activating sensory nerves through actions on ion channels on their peripheral terminals.

Effects on synovitis Synovitis is an integral part of OA pathogenesis. Multinucleated giant cells have been reported in synovitis, these cells are targets for bisphosphonates as are osteoclasts, and may be responsible for the positive effects noted in synovitis. Indeed bisphosphonates have been shown to inhibit macrophage activation in the synovium and reduce synovitis Effects on Bone marrow lesions The formation of bone marrow edema (BME, Bone marrow lesions) is part of OA pathogenesis, and is associated with progressive disease and disability. Several studies have demonstrated that increased remodeling activity in the subchondral region is associated with increased cartilage lesions and the investigators own studies supported by a grant from HSØ (South-East Health Region of Norway), have demonstrated that the presence of increased remodeling activity and vascularization of bone marrow lesions also show association with cartilage degradation. Bisphosphonates may target both the turnover increase, but also angiogenesis as bisphosphonates, and ZA in particular; exert pronounced anti-angiogenic effects.

Direct effects on chondrocytes Chondroprotection with less fibrillation and ulceration has been demonstrated for ZA in an OA models in rabbits and dogs and it has been hypothesized that bisphosphonates may exert an anabolic effect on chondrocytes. In humans, several bisphosphonates have been shown to reduce cartilage degradation as reflected in the biomarker CTXII (C-terminal telopeptides of type 2 collagen).

Clinical trials testing bisphosphonates in OA Bisphosphonates have been tested prospectively as treatment modalities in previous human clinical trials with equivocal results. One trial tested the effects of a less potent bisphosphonate (risedronate) with 4 different doses (5 and 15 mg daily, 35 and 50 mg/week) in knee OA. Joint space width in the placebo group decreased non-significantly by 8 mm vs. 4 and 1mm in the 5 and 15 mg groups, respectively and pain scores did not show significant reductions. Furthermore, serendipitously, the placebo group in the Risedronate trial was very healthy, as it did not exhibit worsening of symptoms over the trial period. This may further have jeopardized the trial outcome. Markers of cartilage degradation, however, revealed significant reductions. In a Japanese study looking at the effects of another oral bisphosphonate, Alendronate, however, Nishii et al. demonstrated significant reductions in VAS and WOMAC pain scores for up to 24 months.

The lack of efficacy of oral bisphosphonates in OA have been primarily ascribed to their poor absorption resulting in lower Cmax after administration (24). Therefore, more recent trials have focused on iv administration, where Cmax will be much higher. Varenna et al randomized 64 patients with OA and demonstrable BML's on MRI to receive either 4 iv. doses (100 mg per infusion of the bisphosphonate Neridronate or placebo. They demonstrated significant reductions in pain, reduced use of analgesics and improved QoL after 50 days. Similar improvements have been reported 5 weeks after intraarticular administration of the bisphosphonate clodronate. Data from the Osteoarthritis initiative demonstrated that patients treated with the iv bisphosphonate zoledronic acid for osteoporosis revealed significant reduction in OA pain scores for up to 3 years. In a later study, Laslett et al demonstrated significant effects on bone marrow edema size and pain in OA over a 1 year period. The doses given in the intravenous trials have been much higher than in the trials using oral administration.

Rationale for dosage and placebo It seems that the dose required for effect on OA should be higher than that which is used for treatment of osteoporosis shown by Varenna et al. Therefore, in this study the investigators choose to treat with two doses of ZA.

As there is no curable treatment for OA, best standard of care is alleviation through paracetamol, NSAIDs or in some cases opioids. Many patients already use one or more of these when they are referred to surgical evaluation. One of the endpoints of this study is to register use of these medications before and after treatment. Using paracetamol instead of placebo could potentially lead to overuse as it can be bought over the counter. Contraindication to NSAID's is common in the elderly population and could exclude many participants.

Simulating the active phase reaction commonly seen with ZA infusion with an active placebo is difficult. However, administration of prednisolone and NSAID's should minimize symptoms.

The investigators experience Based on the published experience with zoledronic acid in OA, the investigators administered two doses of IV. Zoledronic acid (5 mg) with a 3 month interval to patients with osteoporosis and OA of the hip and knee and demonstrable BML on MRI. The dosing regimen was based on previous studies reporting effects of zoledronic acid on bone marrow edema in transient osteoporosis. The patients achieved significant pain reduction as assessed by VAS within a period of 3 and 6 months. VAS decreased 85% from 6,8 (SD 1,8) at baseline to 1,0(0,9) at month 3 and 0,9(0,9) at month 6 (ANOVA p > 0,001). Among these were 3 patients scheduled for surgery. 80% of the patients have been followed for more than 1 year and still exhibit the same degree of pain reduction and increased mobility.

Risk versus benefits The risks of implant surgery are numerous, including infection, thrombosis, dislocation, fracture and in rare instances death. Therefore, a safe and effective conservative management can save the patient from unnecessary complications. The survivorship of hip implants has improved considerably over the last decades, but younger patients are at risk of needing one or more revisions during their lifetime. Revision surgeries are more prone to complications.

The goal of this treatment is to delay or prevent the need for implant surgery. To participate, patients will delay a possible operation for 12 months. Those that are included in the placebo group will not receive any active treatment and cannot expect any better function other than placebo effect. Patients can withdraw from the study at any time.

Although ZA is not approved for treatment of OA, it is regarded as safe for use in adults. The side effects of ZA are rarely serious. Known side effects such as atypical femur fracture and osteonecrosis of the jawbone is extremely rare (1/10.000-1/100.000). Acute phase reactions are common (30%), but usually mild to moderate and lasts 1-3 days. The symptoms can be alleviated with paracetamol, NSAID's or prednisolone.

Microindentation includes injection of local anesthetics and a needle puncture on the tibial bone. No serious adverse events have been recorded.

Magnetic resonance imaging poses no risks given that the participant has no contraindications to imaging such as metal or electronic implants sensitive to magnetic forces.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80
* Continuous worsening of hip pain with an onset of minimum 3 months
* Hip Pain intensity >40mm on a visual analogue scale (VAS) ranging from 0 (no pain) to 100mm (maximal pain) during weight bearing for the last 7 days
* HHS < 65 (Harris Hip Score)
* Hip OA fulfilling the ACR (American College of Rheumatology) criteria [33]
* Hip MRI scan showing large (>1 cm diameter) Bone Marrow lesions (BMLs)
* Willing and able to consent and comply with the study protocol

Exclusion Criteria:

* eGFR (estimated glomerular filtration rate) < 35 ml/min or hypocalcemia
* Exposure to any treatment affecting bone other than Ca+D ( bisphosphonates, Denosumab teriparatide or continuous treatment of prednisolone)
* Diseases affecting bone and joints (i.e inflammatory joint diseases, osteonecrosis with segmental collapse and deformation, primary bone cancer or known skeletal metastases)
* Severe vitamin D deficiency (S-25(OH)D < 25 nmol/l) has to be supplemented with Ca+D before zoledronic acid infusion
* Ipsilateral knee prosthesis
* Contralateral hip prosthesis
* Women of child bearing potential (WOCBP). Female participants must be in a postmenopausal state or permanent sterile.
* Hypersensitivity or previous allergic reaction to ZA or other bisphosphonates.
* Hypersensitivity or previous allergic reaction to Calcigran Forte (a calcium and vitamine D supplement) or Prednisolone

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in joint pain by VAS (Visual analogue pain scale from 1-10) from baseline to 12 months follow up, in the intervention group compared to the placebo group | Baseline and 12 months
  Pain during weight bearing measured with Visual Analogue Pain Scale

SECONDARY OUTCOMES:
Mean change in joint pain by VAS from baseline to 3 and 6 months follow up, in the intervention group compared to the placebo group | baseline, 3 and 6 months
  Pain during weight bearing measured with Visual Analogue Pain Scale
Mean change in function and activity score (HOOS) from baseline to 3, 6 and 12 months follow up, in the intervention group compared to the placebo group | baseline, 3, 6 and 12 months
  Function and activity measured with PROM (patient reported outcome measure) Hip Disability and Osteoarthritis, 0-100 worst to best scale
Mean change in function and activity score (HHS) from baseline to 12 months follow up, in the intervention group compared to the placebo group | 12 months
  Function and activity measured with Harris hips score, 0-100 worst to best score.
Mean change in 40mWT (40 meter walking test measured in seconds) from baseline to 3, 6 and 12 months follow up, in intervention group compared to placebo group | baseline, 3, 6 and 12 months
  40 meter walking test measured in seconds
Mean change in SCT (Stair climb test measured in seconds) from baseline to 3, 6 and 12 months follow up, in intervention group compared to placebo group | baseline, 3, 6 and 12 months
  Stair Climb test measured in seconds (11 stairs)
Mean change in 30CST (Chair stand test, measured by number of repetitions in 30 seconds) from baseline to 3, 6 and 12 months follow up, in intervention group compared to placebo group | baseline, 3, 6 and 12 months
  Chair stand test measured in number of repetitions in 30 seconds
Mean change in QoL (EQ-5D) from baseline to 3, 6 and 12 months follow up, in the intervention group compared to the placebo group | baseline, 3, 6 and 12 months
  Use of Euroqol 5 questions (EQ-5D), measuring disease related quality of life. Score is calculated using value set from English population
Change in mean number of doses of Paracetamol, NSAID and/or opiates per week in each group during the last month compared to baseline at 12 months follow up | baseline, 3, 6 and 12 months
  Change in use of pain medication
Number of AE/SAE (adverse events and serious adverse events) and AR/SAR/SUSAR (adverse/serious adverse and suspected unexpected serious adverse reactions) in the intervention group compared to placebo group 12 months after first infusion. | baseline and 12 months
  Registrating number of adverse effects and adverse reactions

OTHER OUTCOMES:
Change in joint space narrowing (in millimeters) from baseline to 12 months follow up seen on X-ray, compared to the placebo group. | Baseline and 12 months
  exploratory endpoint
Changes in bone turnover in BMLs after treatment with zoledronic acid seen with histomorphometry. A comparison between patients in the treatment and placebo group, that end up with joint implant surgery. | Baseline and 12 months
  Exploratory endpoint. Bone turnover will be assessed after tetracycline double labeling followed by intersection counting of single and double labeled surfaces.
Changes in vascularization in BMLs after treatment with zoledronic acid seen with histomorphometry. A comparison between patients in the treatment and placebo group, that end up with joint implant surgery. | Baseline and 12 months
  Exploratory endpoint. Tissue vascularity will be assessed using point counting.
Changes in bone material properties by impact microindentation (measured in bone material strength index, BMSi) of tibial bone before and after treatment with zoledronic acid compared to the placebo group | Baseline and 12 months
  Exploratory endpoint
Correlation between bone material properties by impact microindentation of tibial bone (BMSi) and Bone turnover markers (BTM)/BML at baseline comparing patient with and without BMLs on hip MRI | Baseline
  Exploratory endpoint
Percentage of participants treated with implant surgery of the affected hip in the treatment group compared to placebo group 12 months after the first infusion. | 12 months
  Exploratory endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Erik F Eriksen, MD, PhD, Study Director — Helse Sor-Ost
Locations (1):
- Martina Hansens Hospital, Sandvika, Norway

IPD SHARING:
Plan to Share IPD: Undecided
No plan has been discussed within the study group yet

REFERENCES:
- [Background] Sellam J, Berenbaum F. The role of synovitis in pathophysiology and clinical symptoms of osteoarthritis. Nat Rev Rheumatol. 2010 Nov;6(11):625-35. doi: 10.1038/nrrheum.2010.159. Epub 2010 Oct 5. PMID 20924410
- [Background] Prieto-Potin I, Largo R, Roman-Blas JA, Herrero-Beaumont G, Walsh DA. Characterization of multinucleated giant cells in synovium and subchondral bone in knee osteoarthritis and rheumatoid arthritis. BMC Musculoskelet Disord. 2015 Aug 27;16:226. doi: 10.1186/s12891-015-0664-5. PMID 26311062
- [Background] Roelofs AJ, Thompson K, Ebetino FH, Rogers MJ, Coxon FP. Bisphosphonates: molecular mechanisms of action and effects on bone cells, monocytes and macrophages. Curr Pharm Des. 2010;16(27):2950-60. doi: 10.2174/138161210793563635. PMID 20722616
- [Background] Moreau M, Rialland P, Pelletier JP, Martel-Pelletier J, Lajeunesse D, Boileau C, Caron J, Frank D, Lussier B, del Castillo JR, Beauchamp G, Gauvin D, Bertaim T, Thibaud D, Troncy E. Tiludronate treatment improves structural changes and symptoms of osteoarthritis in the canine anterior cruciate ligament model. Arthritis Res Ther. 2011 Jun 21;13(3):R98. doi: 10.1186/ar3373. PMID 21693018
- [Background] Khorasani MS, Diko S, Hsia AW, Anderson MJ, Genetos DC, Haudenschild DR, Christiansen BA. Effect of alendronate on post-traumatic osteoarthritis induced by anterior cruciate ligament rupture in mice. Arthritis Res Ther. 2015 Feb 16;17(1):30. doi: 10.1186/s13075-015-0546-0. PMID 25888819
- [Background] Duarte JH. Osteoarthritis: alendronate treatment improves pathology in animal model of OA by blocking osteoclastic bone resorption. Nat Rev Rheumatol. 2014 Aug;10(8):446. doi: 10.1038/nrrheum.2014.107. Epub 2014 Jul 8. No abstract available. PMID 25003767
- [Background] Siebelt M, Waarsing JH, Groen HC, Muller C, Koelewijn SJ, de Blois E, Verhaar JA, de Jong M, Weinans H. Inhibited osteoclastic bone resorption through alendronate treatment in rats reduces severe osteoarthritis progression. Bone. 2014 Sep;66:163-70. doi: 10.1016/j.bone.2014.06.009. Epub 2014 Jun 13. PMID 24933343
- [Background] Permuy M, Guede D, Lopez-Pena M, Munoz F, Gonzalez-Cantalapiedra A, Caeiro JR. Effects of glucosamine and risedronate alone or in combination in an experimental rabbit model of osteoarthritis. BMC Vet Res. 2014 Apr 26;10:97. doi: 10.1186/1746-6148-10-97. PMID 24766775
- [Background] Yu DG, Yu B, Mao YQ, Zhao X, Wang XQ, Ding HF, Cao L, Liu GW, Nie SB, Liu S, Zhu ZA. Efficacy of zoledronic acid in treatment of teoarthritis is dependent on the disease progression stage in rat medial meniscal tear model. Acta Pharmacol Sin. 2012 Jul;33(7):924-34. doi: 10.1038/aps.2012.28. Epub 2012 May 21. PMID 22609837
- [Background] Bagi CM, Berryman E, Zakur DE, Wilkie D, Andresen CJ. Effect of antiresorptive and anabolic bone therapy on development of osteoarthritis in a posttraumatic rat model of OA. Arthritis Res Ther. 2015 Nov 6;17:315. doi: 10.1186/s13075-015-0829-5. PMID 26542671
- [Background] Buckland-Wright JC, Messent EA, Bingham CO 3rd, Ward RJ, Tonkin C. A 2 yr longitudinal radiographic study examining the effect of a bisphosphonate (risedronate) upon subchondral bone loss in osteoarthritic knee patients. Rheumatology (Oxford). 2007 Feb;46(2):257-64. doi: 10.1093/rheumatology/kel213. Epub 2006 Jul 11. PMID 16837470
- [Background] Walsh DA, McWilliams DF, Turley MJ, Dixon MR, Franses RE, Mapp PI, Wilson D. Angiogenesis and nerve growth factor at the osteochondral junction in rheumatoid arthritis and osteoarthritis. Rheumatology (Oxford). 2010 Oct;49(10):1852-61. doi: 10.1093/rheumatology/keq188. Epub 2010 Jun 26. PMID 20581375
- [Background] Yoneda T, Hata K, Nakanishi M, Nagae M, Nagayama T, Wakabayashi H, Nishisho T, Sakurai T, Hiraga T. Involvement of acidic microenvironment in the pathophysiology of cancer-associated bone pain. Bone. 2011 Jan;48(1):100-5. doi: 10.1016/j.bone.2010.07.009. Epub 2010 Jul 14. PMID 20637323
- [Background] Maas O, Joseph GB, Sommer G, Wild D, Kretzschmar M. Association between cartilage degeneration and subchondral bone remodeling in patients with knee osteoarthritis comparing MRI and (99m)Tc-DPD-SPECT/CT. Osteoarthritis Cartilage. 2015 Oct;23(10):1713-20. doi: 10.1016/j.joca.2015.05.014. Epub 2015 May 29. PMID 26028141
- [Background] Shabestari M, Vik J, Reseland JE, Eriksen EF. Bone marrow lesions in hip osteoarthritis are characterized by increased bone turnover and enhanced angiogenesis. Osteoarthritis Cartilage. 2016 Oct;24(10):1745-1752. doi: 10.1016/j.joca.2016.05.009. Epub 2016 May 24. PMID 27233775
- [Background] Tas F, Duranyildiz D, Oguz H, Camlica H, Yasasever V, Topuz E. Effect of zoledronic acid on serum angiogenic factors in patients with bone metastases. Med Oncol. 2008;25(3):346-9. doi: 10.1007/s12032-008-9043-5. Epub 2008 Jan 19. PMID 18204821
- [Background] Wood J, Bonjean K, Ruetz S, Bellahcene A, Devy L, Foidart JM, Castronovo V, Green JR. Novel antiangiogenic effects of the bisphosphonate compound zoledronic acid. J Pharmacol Exp Ther. 2002 Sep;302(3):1055-61. doi: 10.1124/jpet.102.035295. PMID 12183663
- [Background] Lampropoulou-Adamidou K, Dontas I, Stathopoulos IP, Khaldi L, Lelovas P, Vlamis J, Triantafillopoulos IK, Papaioannou NA. Chondroprotective effect of high-dose zoledronic acid: An experimental study in a rabbit model of osteoarthritis. J Orthop Res. 2014 Dec;32(12):1646-51. doi: 10.1002/jor.22712. Epub 2014 Aug 13. PMID 25125266
- [Background] Dearmin MG, Trumble TN, Garcia A, Chambers JN, Budsberg SC. Chondroprotective effects of zoledronic acid on articular cartilage in dogs with experimentally induced osteoarthritis. Am J Vet Res. 2014 Apr;75(4):329-37. doi: 10.2460/ajvr.75.4.329. PMID 24669915
- [Background] Rosa RG, Collavino K, Lakhani A, Delve E, Weber JF, Rosenthal AK, Waldman SD. Clodronate exerts an anabolic effect on articular chondrocytes mediated through the purinergic receptor pathway. Osteoarthritis Cartilage. 2014 Sep;22(9):1327-36. doi: 10.1016/j.joca.2014.07.009. Epub 2014 Jul 17. PMID 25042551
- [Background] Richette P, Roux C. Impact of treatments for osteoporosis on cartilage biomarkers in humans. Osteoporos Int. 2012 Dec;23 Suppl 8:S877-80. doi: 10.1007/s00198-012-2165-9. Epub 2012 Nov 22. PMID 23179570
- [Background] Bingham CO 3rd, Buckland-Wright JC, Garnero P, Cohen SB, Dougados M, Adami S, Clauw DJ, Spector TD, Pelletier JP, Raynauld JP, Strand V, Simon LS, Meyer JM, Cline GA, Beary JF. Risedronate decreases biochemical markers of cartilage degradation but does not decrease symptoms or slow radiographic progression in patients with medial compartment osteoarthritis of the knee: results of the two-year multinational knee osteoarthritis structural arthritis study. Arthritis Rheum. 2006 Nov;54(11):3494-507. doi: 10.1002/art.22160. PMID 17075851
- [Background] Nishii T, Tamura S, Shiomi T, Yoshikawa H, Sugano N. Alendronate treatment for hip osteoarthritis: prospective randomized 2-year trial. Clin Rheumatol. 2013 Dec;32(12):1759-66. doi: 10.1007/s10067-013-2338-8. Epub 2013 Jul 24. PMID 23881439
- [Background] Varenna M, Zucchi F, Failoni S, Becciolini A, Berruto M. Intravenous neridronate in the treatment of acute painful knee osteoarthritis: a randomized controlled study. Rheumatology (Oxford). 2015 Oct;54(10):1826-32. doi: 10.1093/rheumatology/kev123. Epub 2015 May 20. PMID 25998450
- [Background] Varenna M, Zucchi F, Failoni S, Becciolini A, Berruto M. Comment on: Intravenous neridronate in the treatment of acute painful knee osteoarthritis: a randomized controlled study: reply. Rheumatology (Oxford). 2015 Nov;54(11):2117-8. doi: 10.1093/rheumatology/kev302. Epub 2015 Sep 2. No abstract available. PMID 26338662
- [Background] Rossini M, Adami S, Fracassi E, Viapiana O, Orsolini G, Povino MR, Idolazzi L, Gatti D. Effects of intra-articular clodronate in the treatment of knee osteoarthritis: results of a double-blind, randomized placebo-controlled trial. Rheumatol Int. 2015 Feb;35(2):255-63. doi: 10.1007/s00296-014-3100-5. Epub 2014 Aug 1. PMID 25080876
- [Background] Laslett LL, Kingsbury SR, Hensor EM, Bowes MA, Conaghan PG. Effect of bisphosphonate use in patients with symptomatic and radiographic knee osteoarthritis: data from the Osteoarthritis Initiative. Ann Rheum Dis. 2014 May;73(5):824-30. doi: 10.1136/annrheumdis-2012-202989. Epub 2013 Apr 12. PMID 23585518
- [Background] Laslett LL, Dore DA, Quinn SJ, Boon P, Ryan E, Winzenberg TM, Jones G. Zoledronic acid reduces knee pain and bone marrow lesions over 1 year: a randomised controlled trial. Ann Rheum Dis. 2012 Aug;71(8):1322-8. doi: 10.1136/annrheumdis-2011-200970. Epub 2012 Feb 21. PMID 22355040
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Duarte Sosa D, Vilaplana L, Guerri R, Nogues X, Wang-Fagerland M, Diez-Perez A, F Eriksen E. Are the High Hip Fracture Rates Among Norwegian Women Explained by Impaired Bone Material Properties? J Bone Miner Res. 2015 Oct;30(10):1784-9. doi: 10.1002/jbmr.2537. Epub 2015 May 21. PMID 25900016
- [Background] Duarte Sosa D, Fink Eriksen E. Women with previous stress fractures show reduced bone material strength. Acta Orthop. 2016 Dec;87(6):626-631. doi: 10.1080/17453674.2016.1198883. Epub 2016 Jun 20. PMID 27321443
- [Background] Dobson F, Hinman RS, Hall M, Marshall CJ, Sayer T, Anderson C, Newcomb N, Stratford PW, Bennell KL. Reliability and measurement error of the Osteoarthritis Research Society International (OARSI) recommended performance-based tests of physical function in people with hip and knee osteoarthritis. Osteoarthritis Cartilage. 2017 Nov;25(11):1792-1796. doi: 10.1016/j.joca.2017.06.006. Epub 2017 Jun 22. PMID 28647467
- [Background] Altman R, Alarcon G, Appelrouth D, Bloch D, Borenstein D, Brandt K, Brown C, Cooke TD, Daniel W, Feldman D, et al. The American College of Rheumatology criteria for the classification and reporting of osteoarthritis of the hip. Arthritis Rheum. 1991 May;34(5):505-14. doi: 10.1002/art.1780340502. PMID 2025304
- [Background] Miller PD. The kidney and bisphosphonates. Bone. 2011 Jul;49(1):77-81. doi: 10.1016/j.bone.2010.12.024. Epub 2011 Jan 11. PMID 21232648
- [Background] Cipriani C, Pepe J, Clementelli C, Manai R, Colangelo L, Fassino V, Nieddu L, Minisola S. Effect of a single intravenous zoledronic acid administration on biomarkers of acute kidney injury (AKI) in patients with osteoporosis: a pilot study. Br J Clin Pharmacol. 2017 Oct;83(10):2266-2273. doi: 10.1111/bcp.13332. Epub 2017 Jun 27. PMID 28543687
- [Background] Devlin NJ, Shah KK, Feng Y, Mulhern B, van Hout B. Valuing health-related quality of life: An EQ-5D-5L value set for England. Health Econ. 2018 Jan;27(1):7-22. doi: 10.1002/hec.3564. Epub 2017 Aug 22. PMID 28833869
- See also: Video guide to Osteoarthritis Research Society International (OARSI) Physical tests — https://oarsi.org/research/physical-performance-measures